CLINICAL TRIAL: NCT04420637
Title: Impact of the Covid-19 Pandemic on Gastrointestinal and Liver Diseases
Acronym: RetroCov
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: RetroCov
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims primarily

1. to assess the frequency, nature and outcome of liver disease caused or associated with COVD-19 Furthermore, the study also aims
2. to assess the impact of COVID-19 on patients with chronic liver disease or after liver transplantation (frequency of infections, course of disease, outcome)
3. to assess, whether quarantine measures impact on the rate of decompensation of liver cirrhosis
4. to assess whether the intake of antiviral drugs protects against SARS-CoV-2 infection or COVID disease.

DETAILED DESCRIPTION:
The outbreak of the novel coronavirus (SARS-CoV-2)-infected disease (COVID-19) began in Wuhan, Hubei province in December 2019, spread throughout China in early 2020 and developed as a pandemic thereafter. Although the virus mainly causes respiratory symptoms, GI presentations have been reported in and outside of China. Patients may present with anorexia, nausea, vomiting and abdominal discomfort. Also, faecal-oral transmission of the virus is currently discussed. Preliminary, unpublished data from China suggest that patients with GI symptoms may suffer more frequently from severe courses of the disease. Furthermore, liver injury has been observed during COVID-19 disease.

It is currently unclear, whether patients with chronic liver diseases are at a higher risk to contract COVID-19, to develop a more severe disease course or exhibit higher mortality. Preliminary unpublished communications report conflicting data on COVID-19 in patients with chronic liver diseases. According to those reports, it seems that immunosuppressed individuals (e.g. stable patients after liver transplantation or patients with autoimmune liver disease) do not suffer from more severe pulmonary disease when infected with SARS-CoV-2 compared to non-immunosuppressed individuals. To understand the impact of Covid-19 disease on patients with liver diseases, two registries have been launched to collect anonymous data (SECURE-cirrhosis and COVID-Hep.net). As by 1st of April 24 cases with 4 fatalities have been reported, however, this system does not provide enough information to understand the risk of patients in more detail, since it is unknown if all patients are reported and how many patients were at risk. Furthermore, the available data are very superficial.

Besides the direct effects of COVID-19, patients with chronic liver diseases might also be vulnerable to the indirect effects of the pandemic. Quarantine measures may have considerable psychological impact and may cause post-traumatic stress symptoms, confusion, and anger. There is no available data on the impact of quarantine on risk behaviour, such as alcohol consumption or the use of other liver toxic substances. Such behaviour - although destructive for everyone - can increase the risk of decompensation in patients with liver cirrhosis and cause potentially lethal complications which might require intensive care. Furthermore, the difficulty of access to care for patients with chronic diseases may impact negatively on the course of chronic diseases. To date, it is unclear whether the restricted social life and the restrictions in access to care during the pandemic impacts on liver-related morbidity and mortality.

Another possibility of how studying patients with liver diseases can benefit the general population, is to analyse their medications. Patients with chronic liver disease receive a specialised set of drugs, some of which might be effective against SARS-CoV-2. Unfortunately, the first emergency trial using ritonavir/Lopinavir - antiviral substances that are used to treat HIV and HIV/Hepatitis B or C coinfections - showed disappointing results against SARS-CoV-2. However, other antiviral drugs, for example against hepatitis C, could theoretically also be beneficial. It is currently unknown if patients who take drugs against viral hepatitis may be protected against COVID-19 and a retrospective risk assessment might contribute to more informed studies and a more rational distribution of resources.

ELIGIBILITY:
Covid-19 infection treated within the KAGES (Steirische Krankenanstalten GesmBH = Styrian public hospitals)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with Covid-19 infection treated within the hospital group
Sampling Method: Probability Sample
Enrollment: 1366 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
liver disease | through study completion, on average 30 days
  elevated transaminases

SECONDARY OUTCOMES:
COVID infection in patients with chronic liver disease | during the pandemic, at longest until 31.12.2022
  frequency of COVID infection in patients with known chronic liver disease
decompensation of cirrhosis | during the pandemic, at longest until 31.12.2022
  episodes of decompensation of cirrhosis in relation to quarantine measures
Effect of Antiviral drugs on Covid-19 infection | during the pandemic, at longest until 31.12.2022
  frequency of infections in people taking antiviral drugs against hepatitis B or C

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided